CLINICAL TRIAL: NCT05637099
Title: The Value of Repeated Biomarker Measurements During an SBT to Predict Extubation Failure in Mechanically Ventilated ICU Patients
Brief Title: The Value of Repeated BIOMarker Measurements During an SBT to Predict EXtubation Failure in ICU Patients
Acronym: BIOMEXIC
Status: Active, not recruiting | Type: Observational
Sponsor: Henrik Endeman (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor-Investigator, Henrik Endeman, Principal Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL77372.078.21
Record Dates: First submitted 2022-09-07; First posted 2022-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-08

CONDITIONS: Weaning Failure; Mechanical Ventilation; Spontaneous Breathing Trial; Extubation Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Value of Repeated BIOMarker Measurements During an SBT to Predict EXtubation Failure in Mechanically Ventilated ICU Patients

DETAILED DESCRIPTION:
Rationale: In order to prevent extubation failure or unnecessary prolonged ventilation, accurately predicting readiness for extubation is of key importance in ICU care. Currently, clinical criteria and spontaneous breathing trials (SBTs) are used to assess readiness for extubation. Data on the prognostic value of biomarkers in this setting are limited.

Objective: To investigate the association of biomarker measurements (NT-proBNP, hsTroponin-T, CKMB, myoglobin, GDF-15, CRP, IL-6, PCT, Cystatin-C, CA-125, galectin-3, ST-2, albumin) during an SBT with extubation failure in mechanically ventilated ICU patients.

Study design: Multi-centre prospective observational cohort study.

Study population: Adult ICU patients who are mechanically ventilated for more than 48 hours and fulfil readiness-to wean criteria.

Main study parameters/endpoints: Extubation failure (the need for reintubation within 7-days).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study will collect data that is clinically available, but also encompasses repeated biomarker measurements, cardiopulmonary echographic examination and electrocardiography. Because almost all mechanically ventilated ICU patients have an arterial line, blood can be easily sampled without venepuncture and poses negligible risks for the study patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Mechanically ventilated for more than 48 hours
* Fulfilling readiness-to wean criteria
* Written informed consent from the patient or his/her legal representative

Exclusion Criteria:

* Patients with risk factors for laryngeal oedema and a negative cuff leak test (indicating upper airway obstruction with need for steroid treatment)
* Planned replacement of the endotracheal tube for a tracheostomy
* Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICUs of the Erasmus MC, the Franciscus Gasthuis & Vlietland, Groene Hart ziekenhuis, Amphia ziekenhuis, and OLVG, who are mechanically ventilated for more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | 7 days
  The number of patients who were re-intubated within the next 7 days after extubation
All-cause mortality | 7-days
  The number of patients who died within 7 days after extubation

SECONDARY OUTCOMES:
Rescue non-invasive ventilation or high-flow nasal oxygen for post-extubation respiratory insufficiency | 7 days
  The number of patients with rescue non-invasive ventilation or high-flow nasal oxygen for post-extubation respiratory insufficiency
Extubation failure within 48 hours and 72 hours | 48 hours and 72 hours
  The number of patients who re-intubated 48- and 72 hours after extubation
ICU length of stay post-extubation for medical reasons | Up to 1 year
  The length of stay that patients were admitted in the ICU after extubation
ICU re-admission rate within current hospitalization | Up to 1 year
  The number of patients who were readmitted in the ICU within the current hospitalization
All-cause mortality: ICU, hospital, 28-days, 3 and 12 months | 28-days, 3 and 12 months
  The number of patients that died in the ICU, hospital, at 28-days, 3- and 12-months
Major adverse cardiac event | 3 and 12 months
  The number of patients that had a major adverse cardiovascular events (total death, myocardial infarction, coronary revascularization, stroke, and hospitalization because of heart failure or arrhythmia)
Quality of life of patients after ICU and hospital admission | 3 and 12 months
  The quality of life will be measured using the RAND-36 (Units on a scale)
Quality of life of patients after ICU and hospital admission | 3 and 12 months
  The quality of life will be measured using the EQ-5D questionnaire (Units on a scale)

CONTACTS AND LOCATIONS:
Overall Officials: H. Endeman, Dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No